CLINICAL TRIAL: NCT00947648
Title: Are Neutropenic Diets Beneficial to Improve Outcome?
Brief Title: Outpatient Neutropenic Diet Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2008-0369; NCI-2009-01509 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-07-24; First posted 2009-07-28 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-06

CONDITIONS: Leukemia; Neutropenia
Keywords: acute myelogenous leukemia; AML; myelodysplastic syndrome; MDS; Neutropenia; raw fruits and vegetables
MeSH Terms: conditions — Leukemia; Neutropenia; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Vegetables

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- "Raw" Group (Other): Participants will eat cooked food and the addition of raw fruits and vegetables.
  Interventions: Other: Raw Fruits & Vegetables
- "Cooked" Group (Other): Participants will eat only cooked foods.
  Interventions: Other: Cooked Foods

INTERVENTIONS:
Other: Raw Fruits & Vegetables — Diet containing fresh fruits and vegetables in addition to cooked food.
  Arms: "Raw" Group
Other: Cooked Foods — Diet containing only cooked foods.
  Arms: "Cooked" Group

SUMMARY:
The purpose of this study is to evaluate the infection rate of leukemia patients who eat two different diets. Patients in the "raw" group will eat cooked food and the addition of raw fruits and vegetables. Patients in the "cooked" group will eat only cooked foods and this is the standard neutropenic diet with no fresh fruits or vegetables allowed. The primary objective of the study is to evaluate the infection rate of leukemia patients who eat two different diets. The secondary objectives will be the incidence of fever requiring intravenous antibiotics in each group and death rate.

DETAILED DESCRIPTION:
This study is comparing two different diets. The cooked group will be allowed to eat only cooked food and cooked fruits or vegetables. The raw group will be able to eat cooked food and the addition of fresh fruits and vegetables. Patients will be monitored for infection in both groups. There are still certain foods that you are restricted from eating while receiving chemotherapy and you will be given a list of these restrictions.

Study Groups:

If you agree to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups.

Group 1: Raw group: You will be asked to eat at least 1 raw fruit or vegetable every day you are on study.

Group 2: Cooked group: You will eat only cooked foods while on study. The study doctor will give you a list of the foods that you are allowed to eat.

Your medical chart will be monitored while you are on study to check how often you need antibiotics to treat fever. or if you have an infection.

Diet Questionnaire:

You will be asked to fill out a diet questionnaire every week. The questionnaire will have 5 questions about the foods you have been eating. If you have been released from the hospital, you can return the questionnaire during your scheduled hospital visits,which typically take place 3 times per week. You will have no additional visits during this study. The questionnaire should take about 1-2 minutes each time.

Length of Study:

You will be taken off study if your white blood cell count returns to normal. If your white blood cell counts do not return to normal, the maximum time that you may be on study is 6 weeks.

This is an investigational study. There has not been enough research to prove if raw fruits and vegetables can increase your risk of infection. Many hospitals allow neutropenic patients to eat raw fruits and vegetables and other hospitals restrict fresh fruits and vegetables but, this has not been adequately investigated.

Up to 128 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed patients with acute myelogenous leukemia (AML), acute lymphocytic leukemia ( ALL), or myelodysplastic syndrome (MDS) receiving induction chemotherapy or AML, ALL or MDS patients who are in remission receiving consolidation chemotherapy.
2. Patients who will be receiving myelosuppressive chemotherapy for their disease.
3. Patients who will be able to stay in the Houston area for at least 4 weeks.
4. Patients who can speak either English or Spanish.

Exclusion Criteria:

1. Patients who present with an active infection such as pneumonia, bacteremia, urine, c. difficile or cellulitis infection.
2. Patients who are unable to understand the diet questionnaire which will be written in either English or Spanish.
3. Patients who are admitted to the protective environment.
4. Patients who are younger than age 18 will not be entered in the study.
5. Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Number of Bactermia in Each Participant Group | 6 weeks
  Participants evaluated for presence of bacteremia (gram positive, gram negative, and or candidemia). Participants also evaluated for neutropenic fever requiring administration of antibiotics even if the participant does not have a positive blood culture on a weekly basis. At least 2 positive blood cultures are needed for coagulase-negative staphylococci (CoNS) to be considered bacteremia.
Infection Rate | 6 weeks
  Episodes of neutropenic fevers requiring IV antibiotics and or hospitalization because many times patients have an infection but there is no positive blood cultures. Evaluation of bacteremia will be done by the two nurse investigators via a data questionnaire weekly, see Appendix E. Patients will require at least 2 positive blood cultures for coag neg staph to be considered bacteremia and if there are any other questionable organisms that could be a contaminant, an infectious disease expert is one of the co-investigators and this person will be consulted if this positive blood culture is considered an infection. If the patient has a fever requiring antibiotics with this positive blood culture, then this will also be considered as to whether this is a true infection.

CONTACTS AND LOCATIONS:
Overall Officials: Alison E Gardner, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T. M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: U.T. M.D. Anderson Cancer Center Web Site — http://www.ClinicalTrials.org